CLINICAL TRIAL: NCT03775967
Title: Estimation of Sialic Acid and IL10 Levels in Stage 1 and 2 Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Assistant Professor, Ajman University
Other Study IDs: UGD-H-18-10-31-10
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Periodontal Disease
Keywords: sialic acid; IL10; stage 1 periodontal disease; stage 2 periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sialic acid and IL10 are assessed by taking salivary samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sialic acid — sialic acid level estimation in salivary samples
Diagnostic Test: IL10 — IL10 estimation in salivary samples

SUMMARY:
Sialic acid (SA) is the generic term given to a family of acetylated derivatives of neuraminic acid. SA is a 9 carbon monosaccharide. An important function of host SA is to regulate innate immunity. SA is present in several acute phase proteins which are known to be associated with periodontitis. There exists a need for a biomarker, for early detection of disease evolution and more robust therapy efficacy measurements. Till date, there is very little data regarding simultaneous estimation and comparison of total SA content in saliva. IL-10, an anti-inflammatory cytokine, regulates the synthesis of pro-inflammatory cytokines such as IL-1, -2, -6 and stimulates protective antibody production. IL-10 is expressed in both healthy and diseased human periodontal tissues and is reported to be reduced in patients infected with Aggregatibacter actinomycetemcomitans.

The present study was therefore undertaken with an aim, to not only assess the levels of TSA(Total sialic acid levels),but also of IL 10 levels in saliva from stage 1(mild) to stage 2(moderate) periodontitis patients

DETAILED DESCRIPTION:
Selection of patients by grading the patients according to criteria stage 1 and 2 Periodontitis

Obtaining consent from patients participating in the study

Collection of saliva-unstimulated whole saliva, the samples will be stored at -20 degree Centigrade and later placed in a 1.5ml centrifuge tubes which will be placed in a vacuum cool box indicated for laboratory samples and transported to the lab for investigations. It will be centrifuged at 2500 rpm for 10 mins,stored at -80 deg C. SA(sialic acid) levels will be determined by thiobarbutic acid method of aminoff and ELISA methods. SA levels will be measured in mg/dl,IL10 as in direct measurement.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects should be within the age group of 18 to 55 years
* subject should have atleast 18 natural teeth excluding third molars.

Exclusion Criteria:

* History of periodontal debridement or periodontal surgery in preceding six months or any antimicrobial therapy, anti-inflammatory drugs.
* corticosteroids, in previous three months
* systemically compromised individuals
* smokers
* pregnant and lactating women
* Medical history for absence of systemic disorders such as diabetes mellitus
* cardiovascular diseases
* pneumonia
* tuberculosis
* rheumatoid arthritis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients attending the dental clinics in AB Shetty Institute of Dental sciences,Mangalore
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Sialic acid levels in stage 1 periodontitis | From baseline to 3 months
  Sialic acid is measured by taking salivary samples(unstimulated) from stage 1 periodontitis patients
Sialic acid levels in stage 2 periodontitis | From baseline to 3 months
  Sialic acid is measured by taking salivary samples(unstimulated) from stage 2 periodontitis patients
IL10 levels in stage 1 periodontitis | From baseline to 3 months
  IL10 is measured by taking salivary samples(unstimulated) from stage 1 periodontitis patients
IL10 levels in stage 2 periodontitis | From baseline to 3 months
  IL10 is measured by taking salivary samples(unstimulated) from stage 2 periodontitis patients

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty institute of dental sciences, Mangalore, India

IPD SHARING:
Plan to Share IPD: Undecided